CLINICAL TRIAL: NCT01843530
Title: Randomized, Double-blind, Two Arms, Multicenter, Phase III Study of Berinert for Treatment of ACE Induced Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BER-1272-0058-I
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Acute ACE-induced Angioedema
MeSH Terms: interventions — Complement C1 Inhibitor Protein; Cortisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Cortisone, Clemastin + BERINERT
  Interventions: Drug: Berinert; Drug: Clemastin; Drug: Cortisone acetate
- Group 2 (Placebo Comparator): Cortinsone, Clemastin + NaCl
  Interventions: Drug: Clemastin; Drug: Cortisone acetate; Drug: NaCl

INTERVENTIONS:
Drug: Berinert
  Arms: Group 1
Drug: Clemastin
Drug: Cortisone acetate
Drug: NaCl
  Arms: Group 2

SUMMARY:
This trial is a randomized, double-blind, two arms, multicenter, Phase III study of Berinert for treatment of ACE induced Angioedema.

This study should show that Berinert shortens the time to complete resolution of signs and symptoms of acute ACE-induced angioedema of the upper airway tract compared to placebo when given on top of standard treatment. This study should also compare the time to onset of relief as defined by an at least one point reduction on the severity scale of ACE-induced angioedema with Berinert versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study and ability to fulfil all study requirements
* Male or female patients aged >=18 years
* Patients with ACE induced angioedema (grade II-III) with imminent airway obstruction admitted to an Emergency department
* Patient is being treated with ACEi
* Patient must have acute angioedema attack caused by ACEi
* Treatment should be administered within 10 hours after onset of the angioedema
* Patients with angioedema of the head and/or neck (face, lips, cheeks, tongue, soft palate/uvula, pharynx and larynx)
* Male participants and female participants who are not capable of bearing children or who use a method of contraception that is medically approved by the health authority of the respective country
* Signed patient information consent form

Exclusion Criteria:

* Diagnosis of angioedema of other genesis: e.g. hereditary angioedema, C1-inhibitor deficiency, allergic edema, anaphylaxis, insect bite, trauma, abscess, local inflammation, local tumour, post-operative or post-radiogenic edema, salivary gland disorders
* Participation in a clinical study in the past 30 days
* Patients with simultaneous itchiness of skin (acute urticaria)
* Patients with a history of angioedema before taking ACEi
* History of hypersensitivity to any of the study drugs or medicine with a similar chemical structure.
* Pregnancy and/or breastfeeding
* Mental retardation of the patient with restriction of general judgment and awareness
* History of drug abuse (including alcohol and alcoholic liver disorders)
* Potentially unreliable patients
* Patients who are not suitable for the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-11; Primary Completion 2018-10-05 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
time of resolution | 07/2013 until 12/2014
  Berinert shortens the time to complete resolution of signs and symptoms of acute ACE-induced angioedema of the upper airway tract compared to placebo when given on top of standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Bas, Dr., Principal Investigator — Klinikum rechts der Isar
Locations (4):
- Germany (4):
  - Kath. Klinikum Bochum, Med. Klinik III, Bochum
  - Ludwig-Maximilian-Universität, München
  - Klinikum rechts der Isar, Hals-Nasen-Ohren Klinik, München
  - Universitätsklinikum Ulm, HNO, Ulm